CLINICAL TRIAL: NCT04773288
Title: Handy Hygiene of Children: Understanding the Effect of Live Feedback on Handwashing Behavior
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prof. Dr. Thorsten Staake (Other)
Collaborators: University of Turku (Other)
Responsible Party: Sponsor-Investigator, Prof. Dr. Thorsten Staake, Full Professor of Information Systems, University of Bamberg
Organization: Otto-Friedrich-University Bamberg (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: Hand hygiene of children
Record Dates: First submitted 2021-02-09; First posted 2021-02-26 (Actual); Last update posted 2022-02-07 (Actual); Status verified 2022-02

CONDITIONS: Hand Hygiene; Handwashing

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Live feedback provided on display during handwashing (Experimental)
  Interventions: Other: Live feedback during handwashing
- No live feedback provided during handwashing (No Intervention)

INTERVENTIONS:
Other: Live feedback during handwashing — Live feedback provided during handwashing on display
  Arms: Live feedback provided on display during handwashing

SUMMARY:
Objective of the randomized controlled trial is to assess the impact of a digital intervention on hand hygiene of young children. Children in intervention kindergartens / elementary schools will see live instructions and feedback on their current hand washing activity while washing hands. We hypothesize that the digital intervention will improve hand hygiene practices of children in kindergarten / elementary school.

ELIGIBILITY:
Inclusion Criteria:

* children aged between 2 and 7 years of age
* children attending kindergarten

Exclusion Criteria:

* none

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 127 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-07-19 (Actual); Study Completion 2021-07-19 (Actual)

PRIMARY OUTCOMES:
Main effects of live feedback on handwashing of children | Up to 3 months
  Live feedback is hypothesized to change hand washing activities of children in the short- and long-term. Change in hand washing activity is determined with IoT devices measuring water and soap usage (combined into one measure).
Effect of one-time education session on handwashing of children | Up to 1 month
  One-time educational video is hypothesized to change handwashing activity in the short term but declines with time. Change in hand washing activity is determined with IoT devices measuring water and soap usage (combined into one measure).
Habit formation through live feedback on handwashing of children | Up to 3 months
  Hand washing activities of children are hypothesized to remain changed when live feedback is stopped and in locations where no live feedback is available. Change in hand washing activity is determined with questionnaires for children, parents and educators.
Habit formation through live feedback on handwashing of children | Up to 3 months
  Hand washing activities of children are hypothesized to remain changed when live feedback is stopped and in locations where no live feedback is available. Change in hand washing activity is determined with IoT devices measuring water and soap usage (combined into one measure).
Acquisition of competences of children | Up to 3 months
  Live feedback is hypothesized to change competences of children. Change in hand washing activity is determined with questionnaires for children, parents and educators.
Acquisition of competences of children | Up to 3 months
  Live feedback is hypothesized to change competences of children. Change in hand washing activity is determined with IoT devices measuring water and soap usage (combined into one measure).
Self-efficacy of children | Up to 3 months
  Live feedback is hypothesized to change self-efficacy of children. To be measured with questionnaires for children, parents and educators.
Attitude towards technology of parents | Up to 3 months
  Acquisition of competences perceived by parents is hypothesized to be dependent on their attitude towards digital solutions. To be measured with questionnaires for children, parents and educators.

CONTACTS AND LOCATIONS:
Overall Officials: Thorsten Staake, Prof. Dr., Principal Investigator — Otto-Friedrich-University Bamberg; Joanna Graichen, M.Sc., Principal Investigator — Otto-Friedrich-University Bamberg; Carlo Stingl, M.Sc., Principal Investigator — Otto-Friedrich-University Bamberg; Sanna Salanterä, Prof., Principal Investigator — University of Turku; Anni Pakarinen, PhD, Principal Investigator — University of Turku; Riitta Mieronkoski, Principal Investigator — University of Turku
Locations (2):
- University of Turku, Turku, Finland
- Otto-Friedrich-University, Bamberg, Germany